CLINICAL TRIAL: NCT01761734
Title: Pilot Study of Text Message Reminders for Flu Vaccine For Adults
Brief Title: Pilot Text Message for Influenza Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAK5058
Record Dates: First submitted 2012-12-30; First posted 2013-01-07 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Influenza
Keywords: Influenza vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- text message (Experimental): receipt of text message
  Interventions: Behavioral: text message
- usual care (No Intervention): usual care

INTERVENTIONS:
Behavioral: text message
  Arms: text message

SUMMARY:
Influenza is an important and potentially preventable cause of morbidity and mortality, yet only 46% of U.S. adults were vaccinated by the end of the 2011-12 influenza season despite influenza vaccination being widely recommended, effective, and safe. Influenza vaccination rates are even lower in racial/ethnic minority groups. In order to address the problem of low influenza vaccination rates in minority adults, we plan to build on the well-accepted practice of immunization recall-reminders and the emerging practice of using text message to pilot the feasibility of using text messaging to improve influenza vaccination coverage rates in a low health literacy, largely minority, publicly insured adult population.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years of age,
* at least one visit to the AIM clinic during the previous year
* a cell phone number in the registration system
* fluent in English or Spanish. Exclusion criteria

Exclusion Criteria:

* Receipt of influenza vaccination during the 2012-2013 influenza season prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Receipt of an influenza vaccine dose | March 31, 2013
  Proportion of individuals in each group receiving an influenza dose by the end of the influenza season

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University; Steven Shea, MD MS, Principal Investigator — Columbia University; Jessica Singer, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States